CLINICAL TRIAL: NCT02911493
Title: Reducing Sedentary Time in Patients With Heart Failure
Acronym: Rest-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-1330
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Heart Failure
Keywords: sedentary time; number of steps/day; mobility; disability
MeSH Terms: conditions — Heart Failure; Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sedentary Group-Experimental (Experimental): The experimental group will wear an activPAL and have counseling sessions that use the Health Belief Model and Motivational Interviewing strategies to reduce sedentary time.
  Interventions: Behavioral: Reducing Sedentary Behavior
- Physical Activity Group (Active Comparator): The Active Comparative group will wear an activPAL and have counseling sessions that use the Health Belief Model and Motivational Interviewing strategies to increase exercise time.
  Interventions: Behavioral: Physical Activity Group

INTERVENTIONS:
Behavioral: Reducing Sedentary Behavior — The experimental group will wear an activPAL and have counseling sessions that use the Health Belief Model and Motivational Interviewing strategies to reduce sedentary time.
  Arms: Sedentary Group-Experimental
Behavioral: Physical Activity Group — The Active Comparative group will wear an activPAL and have counseling sessions that use the Health Belief Model and Motivational Interviewing strategies to increase exercise time.
  Arms: Physical Activity Group

SUMMARY:
To determine the change in sedentary time and number of steps/day for older patients with heart failure at risk for mobility disability who receive a program to decrease sedentary behavior versus a standard program to increase exercise.

ELIGIBILITY:
Inclusion Criteria:

* NYHA II-IV,
* Age ≥ 65,
* SPPB score of > 4 and ≤ 10 of 12,

  * and deemed (by 1° cardiologist) to be at maximal tolerated dose of heart failure medication (ACE-inhibitor (ACE-I)/angiotensin receptor blocker and beta blocker (BB) for patients with HF with reduced ejection fraction (HFrEF), and
  * blood pressure controlled for HF with preserved ejection fraction (HFpEF) according to the American Heart Failure Association HF guidelines.

Exclusion Criteria:

* Patients requiring medication titration such as ACE-I or BB, (will return to their cardiologist and be eligible after 3 months of stable medication.)
* Oxygen dependent lung disease,
* Orthopedic or neurologic disease that severely limits mobility,
* Active cancer diagnosis except non-melanoma skin cancer,
* Geriatric Depression Scale (GDS) score of ≥ 9 ,
* Limited life-expectancy of <6 months,
* Known dementia or disease that effects ability to learn/follow directions, or
* Failed MiniCog test.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Number of Subjects that are more active than Control. | Monthly for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Boxer, MD, MSc, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado University, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No